CLINICAL TRIAL: NCT03371407
Title: Movement Error-processes and Sensorimotor Adaptation in Parkinsonian Patient
Acronym: Kinarm
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-36; 2016-A01196-45 (Other: ANSM)
Record Dates: First submitted 2017-05-31; First posted 2017-12-13 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Parkinsonian patient under dopaminergic medication
  Interventions: Other: Assessment of behavioral performance and the electrophysiological (EEG) activity in PD patients during the early and more advanced stages of the pathology
- Parkinsonian patient without dopaminergic medication
  Interventions: Other: Assessment of behavioral performance and the electrophysiological (EEG) activity in PD patients during the early and more advanced stages of the pathology
- Control participants
  Interventions: Other: Assessment of behavioral performance and the electrophysiological (EEG) activity in PD patients during the early and more advanced stages of the pathology

INTERVENTIONS:
Other: Assessment of behavioral performance and the electrophysiological (EEG) activity in PD patients during the early and more advanced stages of the pathology — Assessment of behavioral performance and the electrophysiological (EEG) activity in PD patients during the early and more advanced stages of the pathology, using an instrumentation, called the Kinarm, which assess objectively sensory, motor and cognitive functions

SUMMARY:
The aim of the present project is to document the relationship between the behavioral deficits and the electrophysiological anomalies observed in PD patients in tasks involving motor adaptation to visual or mechanical perturbations.

DETAILED DESCRIPTION:
Parkinson Disease (PD) is a neurodegenerative pathology characterized by the death of dopaminergic neurons in of the substantia nigra pars compacta. The main clinical symptoms are akinesia-stiffness-tremor. These motor deficits are due to dysfunction in the network of the basal ganglia that constitute an ensemble of subcortical nuclei involved in movement control and motor learning. The implication of the basal ganglia (BG) in movement sequence learning (i.e. in movement selection processes) has been clearly established. However, their contribution to adaptation of movement execution remains uncertain. Until recently, the vast majority of the studies on motor adaptation have focused on one mechanism in particular: an implicit process through which motor performance is gradually improved on the basis of errors observed in movement execution, recruiting essentially cerebellar loops. Today, a new line of research has emerged seeking to identify different mechanisms contributing to motor adaptation. Specifically, the implication of cognitive strategies and reinforcement learning mechanisms has been the center of several recent studies, which thus have been emphasizing the role of the BG.

The aim of the present project is to document the relationship between the behavioral deficits and the electrophysiological anomalies observed in PD patients in tasks involving motor adaptation to visual or mechanical perturbations. Recent electrophysiological studies have revealed anomalies in the oscillatory activity in the BG-cortex loop in PD; namely the activity in the beta band (~20Hz) presents an excessive synchronization that might contribute to some behavioral symptoms. Interestingly, recent work has demonstrated that the synchronization in the BG and their cortical projections is 1) diminished by treatments such as dopaminergic medication (L-Dopa) or deep brain stimulation of the subthalamic nucleus (NST), and 2) modulated in relation to movement-error processes.

In this project,it is planned to to conduct two studies involving each several studies. The goal of the first study is twofold: first better understand the motor adaptation deficits specific to different stages of PD disease, and then investigate the influence of the dopaminergic medication on the latter. In this purpose, the behavioral performance and the electrophysiological (EEG) activity in PD patients will be examined during the early and more advanced stages of the pathology, on medication or not (ON or OFF L-Dopa). The specific interest of this study in the relationship between the beta-band activity and, on one side, potential deficits in the explicit cognitive strategies recruited in the initial phase of adaptation and, on the other side, anomalies in reinforcement learning mechanisms implicated in motor adaptation. A secondary goal will be to interpret the observations in light of neuroimaging data. The aim of the second study will be to explore oscillatory and synchronized activities in the BG-cortex loops during motor adaptation to visual or mechanical perturbations. The recording of NST LFP and EEG will implicated the participation of implanted PD patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged over 18 years
* Right-handed patients , following the Modified Edinburgh Handedness Inventory
* Patient with Parkinson's disease according to Gibb criteria
* Idiopathic Parkinson's Disease with a history of more than 5 years
* Stimulation electrodes implanted in the 2 subthalamic nuclei in the Functional and Stereotactic Neurosurgery Department of La Timone Hospital (Pr REGIS).
* Dopa-sensitivity greater than 50%
* Absence of signs of cognitive impairment
* Patient who agreed to participate in the study and signed informed consent
* Patient affiliated with a health insurance

Exclusion Criteria:

* Person not likely to participate in the entire study
* Pregnant or likely to be pregnant during the year
* Patients unable to give their informed consent (detainees, adults under guardianship)
* Person unable to understand the nature and purpose of the study, or presneting with understanding difficulties which could compromise the proper conduct of the study
* Person refusing to sign the Informed Consent Form
* A person who is able to give his or her consent but unable to read / write French language
* patient who can not participate in an MRI study according to the criteria listed in the attached form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from Parkinson disease
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-07-04 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
The electrophysiological (EEG) activity by the BioSemi 64 electrodes system | 6 months
  Hertz identification of electrodes where signal fluctuations are the most important.

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Service de Neurologie, Hôpital de la Timone, Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided